CLINICAL TRIAL: NCT06272097
Title: Optimization Program for the Care Management of Wounds With Delayed Healing Risk After Hip Arthroplasty Based on TIME CDST Tool: a Randomized Controlled Trial Protocol
Brief Title: Postoperative Wounds With Delayed Healing Risk of Clinical Trial Registration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danni Feng (Other)
Responsible Party: Sponsor-Investigator, Danni Feng, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201328
Record Dates: First submitted 2024-02-07; First posted 2024-02-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Wound Heal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive an intervention plan based on the TIME CDST tool led by wound specialist nurses at each dressing change.
  Interventions: Behavioral: Intervention program based on TIME-CDST tool led by wound specialist nurses
- Control group (Other): The control group receives a routine wound care program of wound cleaning and dressing changes at each dressing change.
  Interventions: Behavioral: A routine wound care program

INTERVENTIONS:
Behavioral: Intervention program based on TIME-CDST tool led by wound specialist nurses — Based on the TIME CDST tool led by wound specialist nurses, which includes the following five areas: A. Assess patient, well-being and wound; B. Bring in multidisciplinary team and informal carers to promote holistic patient care; C. Control or treat underlying causes and barriers to wound healing; D. Decide appropriate treatment; E. Evaluate and reassess the treatment and wound management outcomes; Give patients health education on wound care management.
  Arms: Intervention group
Behavioral: A routine wound care program — A routine wound care program of wound cleaning and dressing changes
  Arms: Control group

SUMMARY:
this study aims to optimize the components of TIME CDST based on clinical practice and apply the optimized elements to the management of wounds with delayed healing risk after hip arthroplasty to identify and design the key steps in the clinical application of TIME CDST. Through a randomized controlled trial approach, the investigators will conduct a rigorous comparative analysis of the experimental group and the control group. The intervention group will receive an intervention plan based on the TIME CDST tool led by wound specialist nurses at each dressing change, while the control group receive a routine wound care program of wound cleaning and dressing changes at each dressing change. The main research objective is to evaluate the superiority of the experimental group compared with the control group in terms of wound healing time, healing quality, and patient satisfaction. Through the implementation of this study, the investigators expect to provide an effective optimization scheme for the management of postoperative wounds with delayed healing risk in clinical practice, thereby improving patient outcomes and quality of life.

DETAILED DESCRIPTION:
1. Research Background and Objectives Orthopedic surgical wounds present more complex healing challenges compared to other surgical wounds. Hip arthroplasty is the most common type of orthopedic surgery. Due to surgical complexity or patient-specific factors, this procedure is particularly prone to surgical complications such as surgical site infection, wound dehiscence, tissue necrosis, and hematoma, thereby increasing the risk of delayed wound healing postoperatively.To improve the healing outcomes of postoperative wounds with delayed healing, optimizing nursing management protocols is crucial. This study aims to optimize nursing management for wounds with delayed healing risk after hip arthroplasty using the TIME CDST tool and validate its effectiveness.
2. Research Methods Study Design: This study employed a randomized controlled trial design, randomly assigning participants to an experimental group and a control group, which received different nursing management protocols.

   Sample Size: A total of 492 patients are expected to be included, with 246 in the experimental group and 246 in the control group.

   Intervention Measures: Patients in the experimental group will receive nursing management based on the TIME CDST tool, while those in the control group will receive conventional nursing management.

   Evaluation Indicators: The primary outcome measure is wound healing time. Secondary outcome measures include the number of cases with wound healing, wound area reduction rate, ASEPSIS wound scoring system, Stone-Brock Scar Scoring Scale (SBSES), Visual Analog Scale (VAS), patient comfort score, patient satisfaction score, albumin levels, dressing change frequency, and medical costs.Clinical adverse events will be recorded for safety assessment.

   Data collection and analysis: Data will be collected through questionnaire surveys, observation records, statistical analysis, and comparative analysis.
3. Study process Screening and grouping: Patients meeting the inclusion criteria will be screened and randomly assigned to the experimental group and control group.

   Intervention Implementation: The experimental group will receive a nursing management plan based on the TIME CDST tool, while the control group will receive routine nursing management.

   Follow-up and Evaluation: Regularly assess patients' wound conditions, record healing status, and collect patient satisfaction data.

   Data Analysis: Analyze the collected data and compare differences between the experimental group and the control group in terms of various assessment indicators.

   Result Interpretation and Report Writing: Based on the data analysis results, draw conclusions and write the research report.
4. Expected Results

   Through the implementation of this study, the researchers expect to draw the following conclusions:

   The nursing management plan based on the TIME CDST tool can significantly shorten the wound healing time after hip replacement surgery.

   This plan can improve the wound healing rate after hip replacement surgery. This plan can enhance patient satisfaction with nursing services. This plan has practical application and promotion value in clinical practice.
5. Significance and Value of the Study This study holds significant importance and value for optimizing nursing management of wounds with delayed healing risk. Through scientific experimental design and rigorous data analysis, researchers can provide effective nursing management strategies for clinical practice, thereby improving patient outcomes and quality of life. Additionally, the findings of this study can serve as a reference and inspiration for other similar studies, contributing to the advancement and development of the nursing management field.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* First-time recipient of unilateral total HA or hemiarthroplasty;
* Postoperative wound healing delay risk, defined as epithelialization <50% at 2 weeks postoperatively (quantified using a standardized manual planar measurement method: on day 14 postoperatively, a (quantified using a standardized manual planar measurement method: on day 14 postoperatively, a standardized transparent grid membrane with 1mm² graduations is placed vertically over the wound, and the wound perimeter and epithelialization boundary are marked with a surgical marker. boundary are marked with a surgical marker pen; the epithelialized area is defined as pink, non-exudative tissue completely covering the dermis); Normal cognitive and communication abilities;
* Ability to comply with relevant nursing measures;
* Voluntary participation in this trial
* Voluntary participation in this trial and signed informed consent form.

Exclusion Criteria:

* Active infection at the surgical site prior to initial hip surgery; Deep surgical site infection (SSI) or periprosthetic joint infection (PJI) diagnosed or strongly suspected at screening. diagnosed or strongly suspected at screening (based on clinical symptoms, imaging, or aspiration results according to the MSIS/EBJIS criteria);
* Complete wound dehiscence (>2 cm) or exposure of the prosthesis/bone cement, requiring emergency revision surgery;
* Severe vascular insufficiency (ABI <0.5 cm);
* Severe acute and chronic chronic disease (ABI <0.5 cm) insufficiency (ABI <0.6, severe limb ischemia);
* Uncontrolled systemic conditions severely impairing healing potential: severe malnutrition or obesity (BMI≥ 40 kg/m² or≤ 16 kg/m² or serum albumin <2.5 g/dL); Uncontrolled diabetes (HbA1c >9% in the past 3 months); severe heart failure (NYHA IV); severe liver dysfunction (Child-Pugh C); severe renal failure requiring dialysis; active malignant tumors; immunosuppressive therapy (high-dose corticosteroids >10 mg prednisolone); and dose corticosteroids >10 mg prednisone equivalent/day, biologics, or immunosuppressive agents following transplantation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  Wound healing time will be assessed as the primary outcome indicator. Complete epithelialization of the wound is considered as wound healing and the time taken from enrollment to complete wound healing will be recorded for both groups.

SECONDARY OUTCOMES:
Number of cases with wound healing | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  The number of cases in which the wound will be completely epithelialized (defined as pink, non-exudative tissue completely covered by epithelium) during the period from enrollment to the endpoint
The rate of wound area reduction | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  The rate of wound area reduction will be calculated through the following expression: (original wound area - present wound area)/original wound area × 100%. The accuracy of wound area measurements can be improved by placing a uniform wound measuring tape on one side of the wound and taking a picture of the wound area using image processing and analysis with Image J software (National Institutes of Health, Bethesda, MD).
ASEPSIS wound scoring system | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  The ASEPSIS wound scoring system will be used to assess surgical wound infection and healing. This evaluation criteria primarily evaluates multiple aspects including wound characteristics, antibiotic use, wound drainage, local debridement, bacterial culture, hospital stay, and home care of the wound. A higher score indicates more severe wound infection. (Total score: 0 to 10 indicates satisfactory healing; 11 to 20 indicates poor healing; 21 to 30 indicates mild wound infection; 31 to 40 indicates moderate wound infection; and greater than 40 indicates severe wound infection.)
Stony Brook Scar Evaluation Scale (SBSES) | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  The Stony Brook Scar Evaluation Scale (SBSES) will be measured the aesthetic outcome of postoperative wounds, including five criteria: width, height, color, suture line, and overall appearance. Each criterion is scored as 0 or 1, with a total score ranging from 0 (worst) to 5 (best)
The pain intensity | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  The pain intensity is evaluated using the visual analogue scale (VAS). In the absence of pain, a score of 0 represents a painless state; a score of 1 to 3 represents mild pain; a score of 4 to 6 represents moderate pain; and a score of 7 to 10 represents severe pain.
Patient comfort score | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  Use a self-made nursing comfort questionnaire to evaluate the patient's nursing comfort. The questionnaire was conducted on a 10 point scale, with scores>9 indicating extreme comfort, 8-9 indicating relative comfort, 6-7 indicating basic comfort, and<6 indicating discomfort.
Patient satisfaction score | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  Use a self-made nursing satisfaction questionnaire to evaluate the patient's nursing satisfaction. Both questionnaires were conducted on a 10 point scale, with scores>9 indicating very satisfied, 8-9 indicating relative satisfaction, 6-7 indicating basic satisfaction, and<6 indicating dissatisfaction.
Albumin levels | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  Albumin levels
The frequency of dressing changes | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  The frequency of dressing changes
Medical expenses | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  Medical cost expenditure

OTHER OUTCOMES:
Safety evaluation | The time frame is from the date of intervention to the date of complete wound healing or the outcome endpoint, whichever comes first, with an assessment period of 6 months.
  Clinical events were recorded, including reasons for non-healing (infection, hematoma, abscess, wound dehiscence, rejection reaction), antibiotic treatment, readmission, reoperation, amputation, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Danni Feng, Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No